CLINICAL TRIAL: NCT03716453
Title: A Comparative Study of Intraoperative Fentanyl Consumption Guided by Analgesia Nociception Index Versus Standard Protocol in Patients Undergoing Mastectomy
Brief Title: Intraoperative Fentanyl Consumption Guided by Analgesia Nociception Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Thepakorn Sathitkarnmanee, Associate professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HE611339
Record Dates: First submitted 2018-10-21; First posted 2018-10-23 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Postoperative Pain; Postoperative Complications
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications | interventions — AIEOP acute lymphoblastic leukemia protocol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Intraoperative fentanyl administration will be guided by standard protocol
  Interventions: Procedure: Standard protocol
- ANI group (Experimental): Intraoperative fentanyl administration will be guided by ANI protocol
  Interventions: Procedure: ANI protocol

INTERVENTIONS:
Procedure: Standard protocol — Give narcotic according to vital signs
  Arms: Control group
Procedure: ANI protocol — ANI score 50-70 indicates optimal narcotic effect. ANI score > 70 indicated overdosage of narcotic and narcotic should be withheld.
  ANI score < 50 indicates inadequate narcotic and narcotic should be given.
  Arms: ANI group

SUMMARY:
Balanced anesthesia needs optimization of hypnotic, relaxant, and narcotic. Administration of hypnotic drugs can be monitored by bispectral index score (BIS), while the dosage of muscle relaxants can be guided by train-of four (TOF). However, administration of narcotics lacks objective monitor. Overdosage of narcotic may lead to delayed awakening, while underdosage may lead to high degree of postoperative pain. Recently, there is a monitor, Analgesic Nociceptive Index (ANI) monitor, designed to guide the administration of narcotics. There are many descriptive studies supporting the correlation of ANI score and pain score but there are still very few randomized control studies which report the efficacy of ANI in clinical practice.

DETAILED DESCRIPTION:
Objective: To evaluate the efficacy of ANI to guide the administration of intraoperative fentanyl.

Methods: Sixty female patients undergoing breast surgery with balanced anesthesia will be randomized into 2 groups. The first group will receive fentanyl according to standard practice of attending anesthesiologists. The second group will receive fentanyl according to ANI score protocol.

Primary outcome: Postoperative pain numeric rating scale (NRS) score during 60 minutes in postanesthetic care unit (PACU).

Secondary outcomes: Total intraoperative dose of fentanyl and postoperative nausea/vomiting and sedation score in PACU.

ELIGIBILITY:
Inclusion Criteria:

* Adults female undergoing elective breast surgery
* American Society of Anesthesiologists (ASA) classification I-III
* Body mass index (BMI) 18.5-35 kg/m2

Exclusion Criteria:

* Implanted pacemaker
* Cardiac arrythmia
* Autonomic nervous system (ANS) disorder, e.g. epilepsy, stroke
* Chronic opioid use
* Chronic pain
* On beta-blocker, calcium channel blocker, or other drugs to control arrythmia
* Previous mastectomy
* Pregnancy
* On Nsaids

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pain: NRS | during 60 minutes in PACU
  Measure pain numeric rating scale (NRS) every 15 minutes. NRS has a range from 0 to 10 with 0 indicates no pain while 10 indicates worst pain. NRS of 0-3 is mild, 4-6 is moderate, and 7-10 is severe pain.

SECONDARY OUTCOMES:
Intraoperative fentanyl consumption | During intraoperative period
  Cumulative fentanyl used intraoperatively of both groups
Intraoperative ANI score | During intraoperative period
  Intraoperative ANI score of both groups. ANI has a range from 0 to 100 with 0 indicates worst pain while 100 indicates no pain. ANI 0-49 suggests that more opioid is needed. ANI 50-70 indicate optimal analgesic and no opioid is needed. ANI > 70 indicates excessive effect of opioid and opioid should be withheld.
Postoperative nausea/vomiting | During 24 hours postoperatively
  Nausea/vomiting score (PONV score) every 4 hours. PONV score has a range of 0 to 3. N/V scores 0= none, 1= mild, 2= moderate, and 3= severe PONV.
Postoperative sedation score | During 24 hours postoperatively
  Sedation score every 4 hours. Sedation score has a range of 0 to 3 with 0= fully alert, 1= mild sedation, easy to rouse, 2= moderate sedation, arousable with gentle shaking, and 3= deep sedation, not aroused by speaking or gentle shaking.

CONTACTS AND LOCATIONS:
Overall Officials: Sirirat Tribuddharat, MD, PhD, Principal Investigator — Faculty of Medicine, Khon Kaen University
Locations (1):
- Srinagarind Hospital, Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boselli E, Bouvet L, Begou G, Dabouz R, Davidson J, Deloste JY, Rahali N, Zadam A, Allaouchiche B. Prediction of immediate postoperative pain using the analgesia/nociception index: a prospective observational study. Br J Anaesth. 2014 Apr;112(4):715-21. doi: 10.1093/bja/aet407. Epub 2013 Dec 8. PMID 24322571
- [Result] Daccache G, Jeanne M, Fletcher D. The Analgesia Nociception Index: Tailoring Opioid Administration. Anesth Analg. 2017 Jul;125(1):15-17. doi: 10.1213/ANE.0000000000002145. No abstract available. PMID 28628575
- [Result] Dundar N, Kus A, Gurkan Y, Toker K, Solak M. Analgesia nociception index (ani) monitoring in patients with thoracic paravertebral block: a randomized controlled study. J Clin Monit Comput. 2018 Jun;32(3):481-486. doi: 10.1007/s10877-017-0036-9. Epub 2017 Jun 19. PMID 28631050
- [Derived] Tribuddharat S, Sathitkarnmanee T, Sukhong P, Thananun M, Promkhote P, Nonlhaopol D. Comparative study of analgesia nociception index (ANI) vs. standard pharmacokinetic pattern for guiding intraoperative fentanyl administration among mastectomy patients. BMC Anesthesiol. 2021 Feb 13;21(1):50. doi: 10.1186/s12871-021-01272-2. PMID 33581721